CLINICAL TRIAL: NCT05643651
Title: Rivaroxaban Versus Warfarin for Thromboprophylaxis in Children Aged Over 2 Years With Giant Coronary Artery Aneurysms After Kawasaki Disease: a Multicenter, Open-label, Parallel, Exploratory, Randomized Controlled Trial
Brief Title: Rivaroxaban for Children Aged Over 2 Years With Giant Coronary Artery Aneurysms After Kawasaki Disease
Acronym: RIVA-KG
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-399
Record Dates: First submitted 2022-11-25; First posted 2022-12-09 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Kawasaki Disease; Coronary Artery Aneurysm
Keywords: Kawasaki disease; Giant coronary artery aneurysm; Rivaroxaban; Warfarin; Anticoagulation
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome; Coronary Aneurysm | interventions — Rivaroxaban; Aspirin; Clopidogrel; Warfarin; acarboxyprothrombin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Investigator, Participant and Care provider will not be masked. However, sonographer who is responsible for assessing coronary artery lesions should be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban+Antiplatelet drug (Experimental): Rivaroxaban as anticoagulant will be administered with antiplatelet drug for 3 months. Antiplatelet drug can choose Aspirin or Clopidogrel depending on participant medical history and physician's recommendation.
  Interventions: Drug: Rivaroxaban Oral Tablet [Xarelto]; Drug: Aspirin or Clopidogrel
- Standard antithrombotic care (Active Comparator): Warfarin as anticoagulant will be administered with antiplatelet drug for 3 months. Antiplatelet drug can choose Aspirin or Clopidogrel depending on participant medical history and physician's recommendation. International normalized ratio(INR) should be tested once a month and maintained in target range(1.5~2.5).
  2.Aspirin[3 ~5mg/(kg·d), once daily] or Clopidogrel[ 1.0 mg/kg; once daily] according to experienced clinician recommendation and individual condition.
  Interventions: Drug: Aspirin or Clopidogrel; Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban Oral Tablet [Xarelto] — Administered in an age- and bodyweight-adjusted, 15 mg-equivalent dose regimen proposed by model- and clinical evidence-informed precision dosing
  Other Names: Xarelto
  Arms: Rivaroxaban+Antiplatelet drug
Drug: Aspirin or Clopidogrel — Aspirin [3 ~5mg/(kg·d) once daily] or Clopidogrel [1.0 mg/kg; once daily]
  Other Names: Antiplatelet therapy
Drug: Warfarin — Warfarin 0.05~0.12 mg/(kg·d) once daily. INR should maintain within 1.5 to 2.5
  Other Names: Vitamin K Antagonist
  Arms: Standard antithrombotic care

SUMMARY:
Based on population pharmacokinetic model-based simulation, a 15 mg-equivalent, age-, and bodyweight-adjusted dosing regimen for Chinese children with giant coronary artery aneurysms after acute Kawasaki disease was proposed. This exploratory trial aims to evaluate the feasibility, safety and effectiveness of rivaroxaban compared to warfarin for thromboprophylaxis in children aged over 2 years with giant coronary artery aneurysms after Kawasaki disease

DETAILED DESCRIPTION:
Lifelong anticoagulant treatment is required in children with giant coronary artery aneurysm after Kawasaki disease, imposing social and psychologic burdens on patients and parents. Rivaroxaban is a potential oral anticoagulant in this population. Considering the impact of ethnic difference and growth development, we proposed a Chinese-specific, optimized dosing regimen based on model- and clinical evidence-informed precision dosing. In the previous pilot study, this optimized dosing regimen demonstrated a favorable feasibility among 11 Chinese pediatric patients aged over 2 years with giant coronary artery aneurysm after Kawasaki disease, with no thrombosis or major bleeding over 6 months.

This study is a multicenter, open-label, exploratory, randomized controlled trial to evaluate the feasibility, safety and effectiveness of rivaroxaban for thromboprophylaxis in children aged over 2 years with giant coronary artery aneurysms after Kawasaki disease, following the 15 mg-equivalent dosing regimen. Participants will be randomly assigned to the control or experimental groups. Randomization ratio will be 2:1. The control group will receive warfarin plus aspirin or clopidogrel, and the experimental group will receive rivaroxaban plus aspirin or clopidogrel. Baseline characteristics, treatment effect outcomes, bleeding events, adverse events and compliance of intervention of each participant will be collected.

Because this is an exploratory study and the low incidence of giant coronary artery aneurysm in children with Kawasaki disease, the study plans to recruit 100 participants. The aims include:

* The feasibility
* The safety and efficacy profile of the optimized, 15 mg-equivalent dosing regimen
* The group differences in safety and treatment effect between warfarin and rivaroxaban

ELIGIBILITY:
Inclusion Criteria:

1. Giant coronary artery aneurysm(s) in any coronary artery after acute stage of Kawasaki disease. Giant coronary artery aneurysm(s) should be confirmed by two-dimensional echocardiography and meet the diagnostic criteria of Z-score ≥10 or coronary artery internal diameter ≥8mm;
2. Anticoagulant with antiplatelet drug therapy for anti-thromboprophylaxis is recommended for the next 3 months;
3. Participant should be able to tolerate oral feeding, nasogastric or gastric feeding;
4. Children aged ≥ 2 years

Exclusion Criteria:

1. Active bleeding or bleeding risk contraindicating anticoagulant therapy
2. With history of venous thromboembolism or risk factors related with venous thromboembolism, like congenital heart disease, carcinoma, central venous catheter or long-term immobilization.
3. Thrombus within giant coronary aneurysm was confirmed by previous imaging examinations, including two-dimensional echocardiography, computed tomography angiography in coronary artery or coronary angiography
4. An eGFR <30mL/min/1.73 m2 (For children younger than 1 year, serum creatinine results above 97.5th percentile)
5. Platelet count < 100 x 109/L
6. Hepatic disease which is associated with either: coagulopathy leading to a clinically relevant bleeding risk, or alanine aminotransferase > 5x ULN or total bilirubin > 2x ULN with direct bilirubin > 20% of the total
7. Sustained uncontrolled hypertension defined as systolic and/or diastolic blood pressure >95 th age percentile
8. Concomitant use of strong inhibitors of both CYP3A4 and P-glycoprotein, including but not limited to all human immunodeficiency virus protease inhibitors and the following azole-antimycotics agents: ketoconazole, itraconazole, voriconazole, posaconazole, if used systemically (fluconazole is allowed)
9. Concomitant use of strong inducers of CYP3A4, including but not limited to rifampicin, rifabutin, phenobarbital, phenytoin and carbamazepine
10. Hypersensitivity or any other contraindications listed in the local labeling for the comparator treatment or experimental treatment
11. Inability to cooperate with the study procedures and follow-up visits
12. Refuse to provide informed consent eGFR, estimated glomerular filtration rate; ULN, upper level of normal; TB, total bilirubin; CYP3A4, cytochrome P450 isoenzyme 3A4

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Composite of new thrombosis in coronary arteries, major bleeding, clinically relevant non-major bleeding event or major adverse cardiovascular event | From Day 1 of treatment to the third month after treatment initiation
  It is a binary variable. This composite outcome indicates whether any of the following events occurred within 3 months after treatment initiation: (a) newly developed coronary artery thrombosis; (b) major bleeding event; (c) clinically relevant non-major bleeding event; or (d) major adverse cardiovascular event (defined as unstable angina, acute myocardial infarction, hospitalization for heart failure, unplanned coronary revascularization, stroke, or cardiovascular death).

SECONDARY OUTCOMES:
Occurrence of new thrombosis in coronary arteries | From Day 1 of treatment to the third month after treatment initiation
  It is binary data. Every echocardiography conducted during study period will be assessed by masked sonographer. The masked sonographers will assess whether new thrombosis occurs in coronary arteries, and recorded the number of involved coronary arteries.
Time to first new thrombosis in coronary arteries | From Day 1 of treatment to the third month after treatment initiation
  It is time to event data. Every echocardiography conducted during study period will be assessed by masked sonographer. The masked sonographers will assess whether new thrombosis occurs in coronary arteries, and recorded the time to first new thrombosis in coronary arteries.
Composite of Major bleeding or Clinically relevant non-major bleeding event | From Day 1 of treatment to the third month after treatment initiation
  It is a binary variable. Major bleeding is defined as 1.Fatal bleeding; 2.Clinically overt bleeding associated with a decrease in Hgb of ≥20 g/L (2 g/dL) in a 24-h period; 3.Critical site bleeding, such as retroperitoneal, pulmonary, pericardial, intracranial, or otherwise involves the central nervous system; 4.Bleeding that requires an intervention via an invasive procedure; 5.Overt bleeding for which a reversal agent is administered.
  Clinically relevant non-major bleeding event is defined as 1.Bleeding that results in a medical or procedural intervention not meeting major bleeding criteria, including a medication change (reducing, holding, or changing anticoagulation or addition of new medication) ; 2.Bleeding that results in hospitalization or increased level of care; 3.Overt bleeding for which a blood product is administered, and does not meet the criteria for major bleeding
Occurrence of major bleeding | From Day 1 of treatment to the third month after treatment initiation
  It is a binary variable. Major bleeding is defined as 1.Fatal bleeding; 2.Clinically overt bleeding associated with a decrease in Hgb of ≥20 g/L (2 g/dL) in a 24-h period; 3.Critical site bleeding, such as retroperitoneal, pulmonary, pericardial, intracranial, or otherwise involves the central nervous system; 4.Bleeding that requires an intervention via an invasive procedure; 5.Overt bleeding for which a reversal agent is administered.
Occurrence of clinically relevant non-major bleeding (CRNM) | From Day 1 of treatment to the third month after treatment initiation
  It is a binary variable. Clinically relevant non-major bleeding event is defined as 1.Bleeding that results in a medical or procedural intervention not meeting major bleeding criteria, including a medication change (reducing, holding, or changing anticoagulation or addition of new medication) ; 2.Bleeding that results in hospitalization or increased level of care; 3.Overt bleeding for which a blood product is administered, and does not meet the criteria for major bleeding
Occurence of patient important bleeding, no intervention (PIBNI) | From Day 1 of treatment to the third month after treatment initiation
  It is a binary variable. PIBNI is defined as bleeding for which medical attention is sought (phone call, telehealth, clinic, or emergency department visit) but does not result in hospitalization, increased level of inpatient care, or an intervention by the medical team
Occurence of minor bleeding | From Day 1 of treatment to the third month after treatment initiation
  It is a binary variable. Minor bleeding is defined as any overt or macroscopic evidence of bleeding that does not ful ll the above criteria for either fi major bleeding, clinically relevant, non-major bleeding, or patient important bleeding without intervention
Occurrence of major adverse cardiovascular event | From Day 1 of treatment to the third month after treatment initiation
  It is binary variable. Major adverse cardiovascular event (MACE) includes unstable angina, acute myocardial infarction, stroke, hospitalization for heart failure, unplanned revascularization, cardiovascular death. If any of the MACEs occur during the study period, it will be recorded as 1; otherwise, it will be recorded as 0. The definition of each MACE refers to the following guidelines and consensus: 2017 Cardiovascular and Stroke Endpoint Definitions for Clinical Trials, 2019 European society of Cardiology (ESC) guidelines for the diagnosis and management of chronic coronary syndromes, Fourth universal definition of myocardial infarction, and 2023 ESC Guidelines for the management of acute coronary syndromes.
Time to major adverse cardiovascular event | From Day 1 of treatment to the third month after treatment initiation
  It is time to event data. Major adverse cardiovascular event (MACE) includes unstable angina, acute myocardial infarction, stroke, hospitalization for heart failure, unplanned revascularization, cardiovascular death. If any of the MACEs occur during the study period, the time to MACE will be recorded.
Any adverse events | From Day 1 of treatment to the third month after treatment initiation
  It is a text variable. If any adverse events( including durg allergy, severe infection, hepatic dysfunction, renal dysfunction, hypertension, fatigue, abdominal pain or others) occur will be reported to the data and safety monitoring board. The detail of adverse event will be recorded, including classification of adverse event, time of occurrence, symptoms, treatment, resolution time, and outcome.
Plasma concentration of rivaroxaban at specific timepoints | From Day 1 of treatment to the third month after treatment initiation
  For experimental group, plasma concentration of rivaroxaban concentration will be measured by high performance liquid chromatography tandem mass spectrometer. Based on the principle of sparse sampling, predefined timepoints for measurement include: 1. Day 1, 20 minutes -1 h after the first dose; 2. Day 1, 7±1 h after the first dose; 3. After at least three continuous doses (≥ Day 4): before the scheduled dose at that day, which is defined as the trough concentration; 4. After at least three continuous doses (≥ Day 4): 3±1 h the scheduled dose at that day, which is defined as the peak concentration. 5. Peak concentrations during scheduled follow-up: 45±10 days, and 90±10 days; 6. Trough concentrations during scheduled follow-up: 45±10 days, and 90±10 days;
Anti-factor Xa activity at specific timepoints | From Day 1 of treatment to the third month after treatment initiation
  For experimental group, anti-factor Xa activity will be measured by rivaroxaban calibrated chromogenic anti-factor Xa assay. Based on the principle of sparse sampling, predefined timepoints for measurement include: 1. Peak concentrations in scheduled follow-up (45±10 days, and 90±10 days): 3±1 h the scheduled dose at that day; 2. Trough concentrations in scheduled follow-up (45±10 days, and 90±10 days): before the scheduled dose at that day
Discontinuation anticoagulant due to regression of coronary artery lesions | From Day 1 of treatment to the third month after treatment initiation
  It is a binary variable. During study period, researchers will assess and recommend to discontinue anticoagulant if coronary artery lesions regress, which will be confirmed by echocardiography, coronary artery computerized tomography angiography, or coronary artery angiography.
Changes in Z-score of each coronary artery aneurysms | From Day 1 of treatment to the third month after treatment initiation
  This is a repeated measurement. On day 0, an initial echocardiography will be performed by masked sonographer to assess coronary artery lesions. The maximum internal diameter of coronary artery lesion will be measured and recorded. With data of height, bodyweight and internal diameter, Z-score will be calculated (Journal of the American Society of Echocardiography, 2011, 24(1)). If multiple coronary artery aneurysms exists, internal diameter and Z-score will be measured, calculated and recorded separately. Repeated echocardiographies will be conducted at each scheduled visit (45±10 days、90±10 days).
Anticoagulation Monitoring-Related Cost | From Day 1 of treatment to the third months after treatment initiation
  Total healthcare resource utilization cost directly related to anticoagulation monitoring. This includes:
  1. Laboratory test costs (e.g., INR testing cost in the control group, calculated as the number of INR tests multiplied by the unit cost per test; anti-Xa activity testing cost in the intervention group, calculated as the number of anti-Xa tests multiplied by the unit cost per test);
  2. Medical service costs (e.g., additional outpatient or emergency visits, medication adjustments, follow-up visits, consultations, and telephone follow-ups due to abnormal INR values).

OTHER OUTCOMES:
Genetic polymorphism | From Day 1 of treatment to the third month after treatment initiation
  For experimental group, the rest blood sample from rivaroxaban plasma concentration measurement will be collected for genetic polymorphisms examination. Genes related to rivaroxaban metabolism and transport will be examined, including CYP3A4, ABCB1, ABCG2, and et.cl CYP3A4: Cytochrome P450 Family 3 Subfamily A Member 4, ABCB1: ATP Binding Cassette Subfamily B Member 1; ABCG2: ATP Binding Cassette Subfamily G Member 2

CONTACTS AND LOCATIONS:
Overall Officials: Fang Liu, MD, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No